CLINICAL TRIAL: NCT06883110
Title: A Single-Center, Open-Label, Non-Inferiority Clinical Study of Angong Niuhuang Pills With Different Bovine Bezoar Formulation Sources in the Treatment of Acute Ischemic Stroke
Brief Title: Angong Niuhuang Pills With Different Bovine Bezoar Formulation Sources in the Treatment of AIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Daishi Tian, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AgNhWinAIS
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Z11020076 group (Experimental): In addition to receiving standard therapy for acute ischemic stroke (AIS), participants were administered Beijing Tongrentang Angong Niuhuang Pills (3g once daily as a single dose) for 7 consecutive days.
  Note: The AIS standard therapy strictly adhered to first-line treatments recommended by the Chinese guidelines for acute cerebral infarction management.
  Interventions: Drug: Z11020076
- Z20063878 group (Experimental): In addition to receiving standard therapy for acute ischemic stroke (AIS), participants were administered Wuhan Jianmin Dapeng Pharmaceutical Co., Ltd. Angong Niuhuang Pills (3g once daily as a single dose) for 7 consecutive days.
  Note: The AIS standard therapy strictly adhered to first-line treatments recommended by the Chinese guidelines for acute cerebral infarction management
  Interventions: Drug: Z20063878
- blank control group (No Intervention): Participants would receive AIS standard therapy strictly adhered to first-line treatments recommended by the Chinese guidelines for acute cerebral infarction management

INTERVENTIONS:
Drug: Z11020076 — Beijing Tongrentang Angong Niuhuang Pills (3g once daily as a single dose) for 7 consecutive days.
  Arms: Z11020076 group
Drug: Z20063878 — Wuhan Jianmin Dapeng Pharmaceutical Co., Ltd. Angong Niuhuang Pills (3g once daily as a single dose) for 7 consecutive days.
  Arms: Z20063878 group

SUMMARY:
This study is a single-center, open-label, controlled clinical trial that prospectively enrolls 100 participants (40 in the Z11020076 group, 40 in the Z20063878 group, and 20 in the blank control group) to collect clinical data, imaging data, and biospecimens over an 84-day follow-up period. The primary objective is to compare the efficacy and safety of Angong Niuhuang Pills from Beijing Tongrentang (Approval No. Z11020076) and Wuhan Jianmin Dapeng Pharmaceutical Co., Ltd. (Approval No. Z20063878) in improving clinical functional outcomes and prognosis in acute ischemic stroke (AIS) patients. The secondary objective is to evaluate the interventional effects of Angong Niuhuang Pills with different bovine bezoar formulation sources on gut microbiota diversity and composition, peripheral blood immune function, and inflammatory status in AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants or their legal guardians must be capable of understanding the study's purpose and risks and provide informed consent.
* Eligible subjects are aged 18-80 years (inclusive) at the time of consent, regardless of gender.
* All individuals of childbearing potential and male participants must use effective contraception during the study and for at least 6 months after the last dose of the investigational treatment. Additionally, participants must refrain from donating sperm or eggs during the study and for at least 6 months post-treatment.
* Inclusion criteria included: confirmed diagnosis of acute ischemic stroke (AIS) with symptom onset ≤48 hours, NIHSS score of 4-20 (with NIHSS category 1a [level of consciousness] ≥1), and exclusion of intracranial hemorrhage confirmed by imaging (CT or MRI).
* Participants must meet traditional Chinese medicine (TCM) diagnostic criteria for stroke (per the Diagnostic and Efficacy Evaluation Standards for Stroke in TCM issued by the State Administration of Traditional Chinese Medicine), including:Primary symptoms: Hemiplegia, altered consciousness, slurred speech or aphasia, sensory disturbance, facial deviation.Secondary symptoms: Headache, dizziness, pupillary abnormalities, dysphagia, gaze deviation, ataxia.Diagnosis requires ≥2 primary symptoms or 1 primary symptom plus ≥2 secondary symptoms. Written informed consent must be obtained.

Exclusion Criteria:

* Hemorrhagic or mixed stroke.
* Severe cardiac, hepatic, or renal dysfunction or malignancy.
* Prior stroke resulting in a baseline modified Rankin Scale (mRS) score >3.
* Use of medications judged by the investigator to significantly affect gut microbiota or immune function (e.g., antibiotics, immunosuppressants) during the window period (3 days before baseline to 14±3 days post-treatment).
* Allergy to the investigational product or its components.
* Prior participation in this study.
* Blood donation (≥1 unit) within 90 days, plasma donation within 1 week, or platelet donation within 6 weeks before screening.
* Pregnancy, lactation, or plans for pregnancy/breastfeeding during the study or within 30 days post-treatment.
* Concurrent or recent (within 90 days) participation in other clinical trials.
* Clinically significant suicidal ideation or behavior within the past 12 months per Columbia-Suicide Severity Rating Scale (C-SSRS).
* Inability or unwillingness to comply with protocol requirements.
* Significant hearing/visual impairment, language barriers, claustrophobia, or other conditions interfering with neuropsychological assessments or MRI.
* Any other unspecified reasons deemed by the investigator to disqualify participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Score | Day 1, Day 7 (±1), Day 14 (±3), and Day 84 (±5)
NIHSS | Day 1, Day 7 (±1), Day 14 (±3), and Day 84 (±5)
1a score in NIHSS | Day 1, Day 7 (±1), Day 14 (±3), and Day 84 (±5)

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No